CLINICAL TRIAL: NCT04259879
Title: Evaluation of p21 Induction and Molecular Pathways Related to Short-term Fasting Response
Brief Title: Molecular Pathways Related to Short-term Fasting Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IMDEA Food (Other)
Collaborators: Centro Nacional de Investigaciones Oncologicas CARLOS III (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IMD PI0025
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-01

CONDITIONS: Fasting
Keywords: Short-term Fasting; molecular mechanisms; p21; Peripheral blood mononuclear cells (PBMCs); PPARalpha
MeSH Terms: conditions — Fasting; Intermittent Fasting | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Intervention Model Description: This study was an Interventional study. There were three evaluations: the basal one was an initial evaluation after overnight fasting, the second evaluation 24 hours later (36 hours fasting) and the third one 24 hours post-refeeding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fasting (Experimental): The participants will follow a short-term fasting period for 36 hours
  Interventions: Other: Fasting

INTERVENTIONS:
Other: Fasting — Food intake restriction

SUMMARY:
This study will evaluate the effect of short-term fasting (36 hours) in gene expression in blood cells in healthy volunteers.

DETAILED DESCRIPTION:
Fasting is a nutritional intervention consisting on the restriction of nutrient intake during a relatively long period of time. It elicits a profound metabolic reprogramming aimed at shifting nutrient supply from external food intake to internal stored nutrients. Periodic activation of this complex response, termed periodic or intermittent fasting (IF), elicits numerous protective effects against aging, metabolic alterations, neurological disorders and cardiovascular health. Short-term fasting is protective in different stress scenarios, including ischemia reperfusion, bouts of inflammation and chemotherapy-induced toxicity, and improves the anti-tumor efficacy of chemotherapy. Although the basic physiology of fasting is well known, the molecular mechanisms underlying its beneficial effects are not yet completely understood.

In mammals, the response to short-term fasting (from 12 to 48 hours) in terms of nutrient mobilization through the bloodstream has been extensively studied. Fasting follows sequential phases, during which nutrients are released from different storing depots. First, glucose is released from glycogen stores in the liver and muscle. Upon depletion of glycogen, two fasting mechanisms are activated: fatty acids are exported from the adipose tissue into the bloodstream in the form of free fatty acids (FFAs), reaching the liver where they are used to produce ketone bodies, a process termed ketogenesis. Also, gluconeogenesis is activated in the liver, generating glucose mainly from glycerol (released during lipolysis) and amino acids, that originate mainly from muscle breakdown. All these physiological responses are tightly regulated by hormonal and molecular mechanisms.

At the hormonal level, fasting induces a decrease in blood insulin, leptin and ghrelin, and an increase in glucagon levels, while blood adiponectin remains unchanged. Also, several signal transduction pathways are affected by fasting. PPARalpha, a nuclear receptor of fatty acids, becomes activated by the fasting-mediated increase in blood Free fatty Acids (FFAs) and triggers the expression of many target genes in several tissues, including blood cells. It has been shown that the Cyclin Dependent Kinase (CDK) inhibitor p21 is highly upregulated during short-term fasting in many mouse tissues. Moreover, it is known that p21-null mice are unable to endure normal periods of fasting and that p21 is required for the full activation of PPARa target genes both in vivo and in isolated hepatocytes.

In the current study, the investigators wanted to study for the first time molecular mechanisms of fasting that still remained unexplored, specially the expression induction of p21 and PPARalpha signalling pathway. For this, the investigators analyzed blood samples from healthy volunteers subjected to 36 hours of fasting, to explore gene expression in Peripheral Blood Mononuclear Cells (PBMCs).

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 - 50 years old.
* BMI >20<30
* Adequate education level and comprehension of the clinical study
* Willingness to participate in the study as a volunteer and to provide written consent

Exclusion Criteria:

* BMI <20 (thinness)
* BMI >30 (obesity)
* Abnormal low glucose levels after fasting
* Having donated blood less than 8 weeks before starting the study
* Subjects who report special discomfort after previous periods of short fasting
* Diagnosis of type 2 Diabetes mellitus (insulin-dependent)
* Dyslipidemia under pharmacological treatment
* High blood pressure under pharmacological treatment
* Dementia, neurological disease or reduction of cognitive function
* Severe illness (hepatic disease, renal disease, etc
* Taking medications that could affect the lipid and glycemic profiles (statins, fibrate, diuretics, corticoids, anti-inflammatory, hypoglycemic or insulin) 30 days before the beginning of the study.
* Taking medications or substances for weight loss management (15 days before the beginning of the study)
* Pregnancy or lactation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04-07 (Actual); Primary Completion 2016-05-18 (Actual); Study Completion 2016-06-15 (Actual)

PRIMARY OUTCOMES:
Changes in gene expression in PBMCs after fasting | Baseline, 24 hours and 48 hours later
  Expression analysis of p21, Pyruvate Dehydrogenase Kinase 4 (PDK4), Carnitine palmitoyltransferase 1 (CPT1), Adipophilin (ADFP) and Solute carrier family 25, member 50 (SLC25A50) were performed in a HT-7900 Fast Real time polymerase chain reaction (PCR). Quantifications were made applying the ΔCt method (ΔCt = [Ct of gene of interest - Ct of housekeeping]). The housekeeping genes used for input normalization were β-actin (ACTB) and ribosomal protein lateral stalk subunit P0 (RPLP0).

SECONDARY OUTCOMES:
Changes in Insulin levels in response to fasting | Baseline, 24 hours and 48 hours later
  Insulin levels (International Units per milliliter) were measured with a kit from Abbott Laboratories, by luminescent immunoassay using the Architect instrument from Abbott Laboratories.
Changes in Free Fatty Acids levels in response to fasting | Baseline, 24 hours and 48 hours later
  Free fatty acids levels (moles per milliliter) were evaluated with a kit from Abbott Laboratories, by enzymatic spectrophotometric assays using an Architect instrument from Abbott Laboratories.
Changes ketone bodies in response to fasting | Baseline, 24 hours and 48 hours later
  Ketone bodies concentration (moles per milliliter) will be measured with a kit from Sigma-Aldrich, by an enzymatic spectrophotometric assay using an microplate reader from Thermo Fisher.
Changes in leptin levels in response to fasting | Baseline, 24 hours and 48 hours later
  Leptin levels (nanograms per milliliter) were measured with a kit from Mercodia by a non-competitive automatic ELISA immunoanalysis
Changes in lipid profile in response to fasting | Baseline, 24 hours and 48 hours later
  To evaluate lipid improvements the following measurements were considered: Triacylglycerol, Total Cholesterol, low Density Lipoprotein and High-Density Lipoprotein measured by routine laboratory (CQS, Madrid, Spain) methods.
Subjective evaluation of tolerance to fasting | 36 hours of fasting
  To evaluate the tolerance to fasting, participants will fill in a fasting tolerance test based on the symptoms they feel, this will result in a final score of tolerance to fasting.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo J Fernandez-Marcos, PhD, Principal Investigator — IMDEA Food; Manuel Serrano Marugán, PhD, Principal Investigator — Spanish National Cancer Research Center
Locations (1):
- IMDEA Food, Madrid, Spain

REFERENCES:
- [Background] Antoni R, Johnston KL, Collins AL, Robertson MD. Effects of intermittent fasting on glucose and lipid metabolism. Proc Nutr Soc. 2017 Aug;76(3):361-368. doi: 10.1017/S0029665116002986. Epub 2017 Jan 16. PMID 28091348
- [Background] Arnason TG, Bowen MW, Mansell KD. Effects of intermittent fasting on health markers in those with type 2 diabetes: A pilot study. World J Diabetes. 2017 Apr 15;8(4):154-164. doi: 10.4239/wjd.v8.i4.154. PMID 28465792
- [Background] Gotthardt JD, Verpeut JL, Yeomans BL, Yang JA, Yasrebi A, Roepke TA, Bello NT. Intermittent Fasting Promotes Fat Loss With Lean Mass Retention, Increased Hypothalamic Norepinephrine Content, and Increased Neuropeptide Y Gene Expression in Diet-Induced Obese Male Mice. Endocrinology. 2016 Feb;157(2):679-91. doi: 10.1210/en.2015-1622. Epub 2015 Dec 14. PMID 26653760
- [Background] Halberg N, Henriksen M, Soderhamn N, Stallknecht B, Ploug T, Schjerling P, Dela F. Effect of intermittent fasting and refeeding on insulin action in healthy men. J Appl Physiol (1985). 2005 Dec;99(6):2128-36. doi: 10.1152/japplphysiol.00683.2005. Epub 2005 Jul 28. PMID 16051710
- [Background] Mattson MP, Longo VD, Harvie M. Impact of intermittent fasting on health and disease processes. Ageing Res Rev. 2017 Oct;39:46-58. doi: 10.1016/j.arr.2016.10.005. Epub 2016 Oct 31. PMID 27810402
- [Background] Varady KA, Bhutani S, Church EC, Klempel MC. Short-term modified alternate-day fasting: a novel dietary strategy for weight loss and cardioprotection in obese adults. Am J Clin Nutr. 2009 Nov;90(5):1138-43. doi: 10.3945/ajcn.2009.28380. Epub 2009 Sep 30. PMID 19793855
- [Background] Vasconcelos AR, Yshii LM, Viel TA, Buck HS, Mattson MP, Scavone C, Kawamoto EM. Intermittent fasting attenuates lipopolysaccharide-induced neuroinflammation and memory impairment. J Neuroinflammation. 2014 May 6;11:85. doi: 10.1186/1742-2094-11-85. PMID 24886300
- [Background] Tinkum KL, Stemler KM, White LS, Loza AJ, Jeter-Jones S, Michalski BM, Kuzmicki C, Pless R, Stappenbeck TS, Piwnica-Worms D, Piwnica-Worms H. Fasting protects mice from lethal DNA damage by promoting small intestinal epithelial stem cell survival. Proc Natl Acad Sci U S A. 2015 Dec 22;112(51):E7148-54. doi: 10.1073/pnas.1509249112. Epub 2015 Dec 7. PMID 26644583
- [Background] Safdie FM, Dorff T, Quinn D, Fontana L, Wei M, Lee C, Cohen P, Longo VD. Fasting and cancer treatment in humans: A case series report. Aging (Albany NY). 2009 Dec 31;1(12):988-1007. doi: 10.18632/aging.100114. PMID 20157582
- [Background] Raffaghello L, Safdie F, Bianchi G, Dorff T, Fontana L, Longo VD. Fasting and differential chemotherapy protection in patients. Cell Cycle. 2010 Nov 15;9(22):4474-6. doi: 10.4161/cc.9.22.13954. Epub 2010 Nov 15. PMID 21088487
- [Background] Lee C, Raffaghello L, Brandhorst S, Safdie FM, Bianchi G, Martin-Montalvo A, Pistoia V, Wei M, Hwang S, Merlino A, Emionite L, de Cabo R, Longo VD. Fasting cycles retard growth of tumors and sensitize a range of cancer cell types to chemotherapy. Sci Transl Med. 2012 Mar 7;4(124):124ra27. doi: 10.1126/scitranslmed.3003293. Epub 2012 Feb 8. PMID 22323820
- [Background] Di Biase S, Lee C, Brandhorst S, Manes B, Buono R, Cheng CW, Cacciottolo M, Martin-Montalvo A, de Cabo R, Wei M, Morgan TE, Longo VD. Fasting-Mimicking Diet Reduces HO-1 to Promote T Cell-Mediated Tumor Cytotoxicity. Cancer Cell. 2016 Jul 11;30(1):136-146. doi: 10.1016/j.ccell.2016.06.005. PMID 27411588
- [Background] Pietrocola F, Pol J, Vacchelli E, Rao S, Enot DP, Baracco EE, Levesque S, Castoldi F, Jacquelot N, Yamazaki T, Senovilla L, Marino G, Aranda F, Durand S, Sica V, Chery A, Lachkar S, Sigl V, Bloy N, Buque A, Falzoni S, Ryffel B, Apetoh L, Di Virgilio F, Madeo F, Maiuri MC, Zitvogel L, Levine B, Penninger JM, Kroemer G. Caloric Restriction Mimetics Enhance Anticancer Immunosurveillance. Cancer Cell. 2016 Jul 11;30(1):147-160. doi: 10.1016/j.ccell.2016.05.016. PMID 27411589
- [Background] Ruderman NB. Muscle amino acid metabolism and gluconeogenesis. Annu Rev Med. 1975;26:245-58. doi: 10.1146/annurev.me.26.020175.001333. No abstract available. PMID 1096762
- [Background] Cahill GJ Jr, Owen OE, Morgan AP. The consumption of fuels during prolonged starvation. Adv Enzyme Regul. 1968;6:143-50. doi: 10.1016/0065-2571(68)90011-3. No abstract available. PMID 5720334
- [Background] Nuttall FQ, Almokayyad RM, Gannon MC. Comparison of a carbohydrate-free diet vs. fasting on plasma glucose, insulin and glucagon in type 2 diabetes. Metabolism. 2015 Feb;64(2):253-62. doi: 10.1016/j.metabol.2014.10.004. Epub 2014 Oct 8. PMID 25458830
- [Background] Nuttall FQ, Almokayyad RM, Gannon MC. The ghrelin and leptin responses to short-term starvation vs a carbohydrate-free diet in men with type 2 diabetes; a controlled, cross-over design study. Nutr Metab (Lond). 2016 Jul 22;13:47. doi: 10.1186/s12986-016-0106-x. eCollection 2016. PMID 27453716
- [Background] Merl V, Peters A, Oltmanns KM, Kern W, Born J, Fehm HL, Schultes B. Serum adiponectin concentrations during a 72-hour fast in over- and normal-weight humans. Int J Obes (Lond). 2005 Aug;29(8):998-1001. doi: 10.1038/sj.ijo.0802971. PMID 15917861
- [Background] Bouwens M, Afman LA, Muller M. Fasting induces changes in peripheral blood mononuclear cell gene expression profiles related to increases in fatty acid beta-oxidation: functional role of peroxisome proliferator activated receptor alpha in human peripheral blood mononuclear cells. Am J Clin Nutr. 2007 Nov;86(5):1515-23. doi: 10.1093/ajcn/86.5.1515. PMID 17991667
- [Background] Lopez-Guadamillas E, Fernandez-Marcos PJ, Pantoja C, Munoz-Martin M, Martinez D, Gomez-Lopez G, Campos-Olivas R, Valverde AM, Serrano M. p21Cip1 plays a critical role in the physiological adaptation to fasting through activation of PPARalpha. Sci Rep. 2016 Oct 10;6:34542. doi: 10.1038/srep34542. PMID 27721423
- [Background] Prokesch A, Graef FA, Madl T, Kahlhofer J, Heidenreich S, Schumann A, Moyschewitz E, Pristoynik P, Blaschitz A, Knauer M, Muenzner M, Bogner-Strauss JG, Dohr G, Schulz TJ, Schupp M. Liver p53 is stabilized upon starvation and required for amino acid catabolism and gluconeogenesis. FASEB J. 2017 Feb;31(2):732-742. doi: 10.1096/fj.201600845R. Epub 2016 Nov 3. PMID 27811061
- [Background] Tinkum KL, White LS, Marpegan L, Herzog E, Piwnica-Worms D, Piwnica-Worms H. Forkhead box O1 (FOXO1) protein, but not p53, contributes to robust induction of p21 expression in fasted mice. J Biol Chem. 2013 Sep 27;288(39):27999-8008. doi: 10.1074/jbc.M113.494328. Epub 2013 Aug 5. PMID 23918930